CLINICAL TRIAL: NCT06376851
Title: DECIDE Registry: AI DErived Plaque Quantification: CCTA and AI-QCPA for Determining Effective CAD Management
Brief Title: AI DErived Plaque Quantification: CCTA and AI-QCPA for Determining Effective CAD Management
Acronym: DECIDE
Status: Active, not recruiting | Type: Observational
Sponsor: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-910-001
Record Dates: First submitted 2024-03-28; First posted 2024-04-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease
Keywords: CAD; AI-QCPA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Group 1: No AI-QCPA: This group includes previously scanned, symptomatic patients with plaque detected and no prior revascularization. No AI-QCPA will be provided.
- Group 2: Delayed AI-QCPA: This group includes previously scanned, symptomatic patients with plaque detected and no prior revascularization. Ninety days following the CCTA, an AI-QCPA report will be provided to the CCTA reader who will in turn provide it to the treating clinician. The treating clinician will decide if changes to medical management are required to effectively treat the patient and if so, treating clinician will contact the patient with the new treatment plan.
  Interventions: Diagnostic Test: AI-enabled quantitative coronary plaque analysis (AI-QCPA)
- Group 3: Stress Test Only: This group includes symptomatic patients who previously had non-invasive stress testing only with no CCTA and no prior revascularization. No AI-QCPA will be provided.
- Group 4: Prospective AI-QCPA, symptomatic without prior revascularization: This group includes newly scanned, symptomatic patients with plaque detected and no prior revascularization. Patients in this group will have current symptoms suggestive of CAD and will not have had prior revascularization. CCTA reader who identifies plaque orders AI-QCPA to inform the medical management plan for the patient.
  Interventions: Diagnostic Test: AI-enabled quantitative coronary plaque analysis (AI-QCPA)
- Group 5: Prospective AI-QCPA, prior PCI: This group includes newly scanned patients with plaque detected. Patients in this group can by symptomatic or asymptomatic and will have had prior PCI in only one vessel territory (CABG patients are not eligible). CCTA reader who identifies plaque orders AI-QCPA to inform the medical management plan for the patient.
  Interventions: Diagnostic Test: AI-enabled quantitative coronary plaque analysis (AI-QCPA)
- Group 6: Prospective AI-QCPA, asymptomatic without prior revascularization: This group includes newly scanned, asymptomatic patients with plaque detected and no prior revascularization. Patients in this group will not have current symptoms suggestive of CAD and will not have had prior revascularization. CCTA reader who identifies plaque orders AI-QCPA to inform the medical management plan for the patient.
  Interventions: Diagnostic Test: AI-enabled quantitative coronary plaque analysis (AI-QCPA)

INTERVENTIONS:
Diagnostic Test: AI-enabled quantitative coronary plaque analysis (AI-QCPA) — The HeartFlow Plaque Analysis provides plaque identification, quantification, and characterization and is meant to support qualified clinicians to aid in the evaluation and risk assessment of coronary artery disease (CAD). It provides data on the volume and type of plaque present (Calcified, Non-calcified, Low Attenuation), both vessel specific and total volumes, with which physicians can better understand a patient's risk, discuss heart health, and help optimize medical management. Plaque Analysis is calculated using image data from a previously acquired CCTA.
  Groups: Group 2: Delayed AI-QCPA; Group 4: Prospective AI-QCPA, symptomatic without prior revascularization; Group 5: Prospective AI-QCPA, prior PCI; Group 6: Prospective AI-QCPA, asymptomatic without prior revascularization

SUMMARY:
The objective of HeartFlow's DECIDE Registry is to collect observational data about the management of patients before and after HeartFlow Artificial Intelligence-Quantitative Coronary Plaque Analysis (AI-QCPA).

DETAILED DESCRIPTION:
The DECIDE Registry is a post-market, multi-center, data collection study assessing the change in management of clinically stable patients who undergo CCTA with plaque detected. Data will be retrospectively collected following the CCTA, and analyses will be completed 90 days, 180 days, and 1 year after CCTA. Data may be retrospectively collected annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria (all must be present) :

1. Groups 1, 2,4,5 and 6: CCTA and plaque detected
2. Group 3: Any patient with a stress test (stress echocardiogram or nuclear imaging including SPECT or PET) and no CCTA within the 90 days prior to site activation
3. Groups 1,2,3 and 4: Clinically stable, symptomatic
4. Group 6: Clinically stable without symptoms suggestive of CAD at the time of the CCTA

Exclusion Criteria (all must be absent) :

1. ED presentation (at the time of the CCTA or stress test)
2. Groups 1,2,3,4, and 6: Previous history of CAD (prior to the CCTA or stress test with history of revascularization)
3. Group 5: Prior history of PCI in multiple vessel territories, PCI in the Left Main, CABG, and/or any other conditions or limitations which would prevent successful CCTA processing by HeartFlow
4. Acute chest pain (in patients who have not been ruled out for ACS)
5. Previously evaluated with and/or in a study which includes AI-QCPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Deidentified data will be collected for all patients who have had a CCTA with plaque detected or a stress test and are included by the site in the registry.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2030-03-27 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 90 Days
  The primary endpoint of the DECIDE Registry is the change in medical management following HeartFlow AI-QCPA at 90 days compared to medical management following CCTA alone. The primary endpoint will only be assessed in patients in Group 2.

SECONDARY OUTCOMES:
Change in LDL levels | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Change in HbA1c levels | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Changes in Non HDL levels | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Changes in HDL levels | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Changes in TG levels | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Changes in weight | From baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups
Reclassification rate of medical management (across the groups) | 90 Days, 180 Days and 365 Days
  Change in preventive medical management (lower or intensify).
Rates of referral to invasive coronary angiography and coronary revascularization (PCI+CABG) | 90 Days, 180 Days and 365 Days
  across the groups
Reclassification rate of symptoms | 90 Days, 180 Days and 365 Days
  Improvement in symptoms across the groups
Number of CV hospitalizations | At 365 Days (and potentially out to 5 years)
  across the groups
Number of Revascularizations | 365 Days
  At one year across the groups

OTHER OUTCOMES:
Number of MACE (CV-related death, MI, or CAD hospitalization) | At 365 Days (and potentially out to 5 years)
  Exploratory & safety endpoints will be compared across the groups unless otherwise noted
Timing of referral to other provider(s) for management | Group 1 vs. Group 2 at 90 days post AI-QCPA and Group 2 vs. 4 at 90 days post AI-QCPA
  across the groups unless otherwise noted
Timing of lab orders (Group 1 vs. Group 2) | Group 1 vs. Group 2 at 90 days post AI-QCPA and Group 2 vs. 4 at 90 days post AI-QCPA
  across the groups unless otherwise noted
Change in Lp(a) (Group 2) | Baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups unless otherwise noted
Change in Lp(a) (Group 4 compared to Group 1) | Baseline to 90 days, from 90 days to 180 days, and 90 days to 365 days
  across the groups unless otherwise noted
Rate of cardiac testing | At 365 Days (and potentially out to 5 years)
  Efficiency of testing based upon imaging and reports for all other cardiac tests including CCTA, SPECT, echo, CAC, and stress echo

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rinehart, MD, Principal Investigator — CAMC Health System; Leslee Shaw, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Moses Cone Memorial Hospital, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No